CLINICAL TRIAL: NCT01337700
Title: Milnacipran in Autism and the Functional Locus Coeruleus and Noradrenergic Model of Autism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Eric Hollander, Clinical Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-09-299
Record Dates: First submitted 2010-12-27; First posted 2011-04-19 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Autism Spectrum Disorder; Asperger Syndrome; Aspergers Syndrome
Keywords: ASD; Autism; Autism Spectrum Disorder; Asperger Syndrome; Asperger; PDD; PDD-NOS
MeSH Terms: conditions — Autism Spectrum Disorder; Asperger Syndrome; Autistic Disorder | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milnacipran (Experimental)
  Interventions: Drug: Milnacipran
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — Patients will receive a titrated dose of milnacipran increasing to a maximum of 100mg a day over the 12 week study period. Dosing will be based on a fixed schedule that will be monitored using a side effect profile.
  Other Names: Savella
  Arms: Milnacipran
Drug: Placebo — Subjects will be given placebo tablets at dosing corresponding to the fixed schedule between 12.5mg and 100mg.
  Arms: Placebo

SUMMARY:
Autism Spectrum Disorders (ASD) include Autistic disorder, Asperger's syndrome and Pervasive Developmental Disorder Not Otherwise Specified (PDD-NOS). These are developmental disorders beginning prior to three years of age. Recent Centers for Disease Control (CDC) estimates suggest that ASD affects up to 1 in 100 individuals and up to 1 in 50 boys. There are very substantial costs associated with caring for patients with ASD, and ASD has the highest Caregiver Burden Scores of any condition. There are three core symptom domains of ASD, including social deficits, repetitive behaviors and language deficits. Patients can also have associated symptoms of attentional deficits, disruptive behaviors and intellectual disability. There is currently no Food and Drug administration (FDA) approved treatment for the core symptoms of autism, but risperidone and aripiprazole have FDA approval for disruptive behaviors associated with autism.

This is a 12 week randomized double blind placebo controlled trial of Milnacipran in adults with ASD or Aspergers Syndrome. Milnacipran is said to play a role in the activation and normalization of the locus coeruleus-noradrenergic system, of which is hypothesized to play a role in behavior adaptations and performance.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients
* Aged 18-50 years
* Diagnosis of Autism Spectrum Disorder
* intelligence quotient greater than 70

Exclusion Criteria:

* Pregnant subjects
* Patients deemed by comprehensive psychiatric interview to have a significant risk of suicide

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, Albert Einstein College of Medicine, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Milnacipran | Placebo
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Milnacipran | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (3.391) | 25.2 (9.149) | 25.10 (6.506)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Severity of Illness [Mean (Full Range); unit: units on a scale] — Scores are using the Clinical Global Impression Scale -Severity (CGI-S). This is a 7-point scale, from 1 (normal not at all ill) to 7 (among the most extremely ill), that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis.
  units on a scale | 4 [4 to 4] | 5 [5 to 5] | 4.5 [4 to 5]
Aberrant Behavior Checklist - Hyperactivity Scale (ABC-H) [Mean (Full Range); unit: units on a scale] — ABC-H can assess problematic behavior at home, in educational and work settings, and in residential and community-based facilities specifically in regard to hyperactivity. It is a sub- scale of the larger ABC-2 which rates 58 specific symptoms, and provides comprehensive descriptions, for each assessed behavior. It is further divided into five sub-scales and the one discussed here is hyperactivity. Each question is rated on a scale from 0-3 with 0 being not problematic and 3 being most problematic.
  units on a scale | 19 [8.45 to 29.55] | 9.8 [3.91 to 15.69] | 14.4 [3.91 to 29.55]
CAARS Inattention/Memory T Score [Mean (Full Range); unit: T score] — The Conners Adult ADHD Rating Scales (CAARS) are the international standard for questionnaire assessment of ADHD. The raw scores are converted to T-scores for each scale and sub-scale which are then compared against the mean. This sub-scale being assessed is inattention/ memory. Higher values represent a worse outcome. A T-score of 50 is the mean of a relevant reference population. A T-score above 65 indicates a moderate to severe problem.
  T score | 68.6 [53.77 to 83.43] | 71.8 [65.99 to 77.6] | 70.2 [53.77 to 83.43]
CAARS Hyperactivity/Restlessness T Score [Mean (Full Range); unit: T score] — The Conners Adult ADHD Rating Scales (CAARS) are the international standard for questionnaire assessment of ADHD. The raw scores are converted to T-scores for each scale and sub-scale which are then compared against the mean. Higher values represent a worse outcome. A T-score of 50 is the mean of a relevant reference population. A T-score above 65 indicates a moderate to severe problem.This sub-scale being assessed is hyperactivity/ restlessness.
  T score | 55 [42.37 to 67.63] | 50.8 [49.24 to 59.56] | 52.9 [42.37 to 67.63]
CAARS Impulsivity/Emotional Labiality T Score [Mean (Full Range); unit: T score] — The Conners Adult ADHD Rating Scales (CAARS) are the international standard for questionnaire assessment of ADHD. The raw scores are converted to T-scores for each scale and sub-scale which are then compared against the mean. Higher values represent a worse outcome. A T-score of 50 is the mean of a relevant reference population. A T-score above 65 indicates a moderate to severe problem.This sub-scale being assessed is impulsivity/ emotional labiality.
  T score | 55.2 [47.54 to 62.86] | 49.2 [43.31 to 55.09] | 52.2 [43.31 to 62.86]

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on Conners Adults Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale
Description: Change will be measured in each subject's score on the Conners Adults Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale from baseline through study end (week 12).Higher values represent a worse outcome.
  The raw scores are converted to T-scores for each scale and sub-scale which are then compared against the mean. Higher values represent a worse outcome. A T-score of 50 is the mean of a relevant reference population. A T-score above 65 indicates a moderate to severe problem. For example, Row 1 is the mean of baseline T-scores for the Inattention/ Memory subscale and Row 2 is the mean of week 12 T-scores for the Inattention/ Memory subscale. The difference between these two means is used to measure the change from baseline through week 12 for both the groups.
Time Frame: Baseline and Week 12 scores
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Milnacipran: Milnacipran: Patients will receive a titrated dose of milnacipran increasing to a maximum of 200mg a day over the 12 week study period. Dosing will be based on a fixed schedule that will be monitored using a side effect profile.
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 5 | 5
T-score
  Baseline: T-SCORES- Inattention/Memory | 68.6 (14.83) | 71.8 (5.81)
  Week 12: T-SCORES- Inattention/Memory | 53.4 (13.05) | 57 (20.22)
  Baseline: T-SCORES- Hyperactivity/Restlessness | 55 (12.63) | 50.8 (8.76)
  Week 12:T-SCORES -Hyperactivity/Restlessness | 44.8 (8.76) | 39.8 (7.56)
  Baseline: T-SCORES- Impulsivity/Emotional Lability | 55.2 (7.66) | 49.2 (5.89)
  Week 12: T-SCORES- Impulsivity/Emotional Lability | 47.8 (6.22) | 43.6 (13.90)

2. Primary Outcome: Change in Hyperactivity as Measured by Aberrant Behavior Checklist - Hyperactivity Scale
Description: The Aberrant Behavior Checklist is an informant-based questionnaire consisting of 58 items subdivided amongst 5 scales: irritability, lethargy and social withdrawal, stereotypic behavior, hyperactivity/non-compliance, and inappropriate speech [34]. A score for each item ranges from 0 indicating "no problem" to 3 indicating "severe problem". Scale scores are calculated by summing the items within that scale. Higher scores indicate greater impairment.Reported Data is for change in ABC-H from baseline to endpoint (week 0 to week 12).This data is specifically looking at the hyperactivity scale which is 16 items with each item ranging from 0-3 making total scores 0-48.
Time Frame: Baseline to Endpoint - 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 5 | 5
units on a scale | -10.4 (12.46) | -4.2 (7.26)

3. Secondary Outcome: Change in Autism Severity Levels Based on the Clinical Global Impressions Scale
Description: The CGI-I reflects the rater's impression of the subject's current autism severity on a 7-point scale ranging from Much Improved (1) to Much worse (5).
Time Frame: screening, baseline, weeks 2,4,6,8,10,12
Measure: Count of Participants; unit: Participants
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 5 | 5
Participants
  Much Improved | 1 | 1
  Minimally Improved | 1 | 1
  No Change | 3 | 2
  Minimally Worse | 0 | 1
  Much Worse | 0 | 0

4. Secondary Outcome: Change in Repetitive Behaviors Using YBOCS-Compulsion and Rigidity Subscale
Description: This scale has been shown to be a sensitive outcome measure in autism trials of repetitive behaviors. Data for secondary outcome not analyzed due to lack of significance in primary outcomes measured.
  * scale range: 0 - 40 total, 0 - 7 subclinical, 8-15 mild, 16 - 23 moderate, 24 - 31 severe, 32 - 40 extreme
  * score interpretation: Higher overall scores reflect increasing symptom severity.
Time Frame: baseline, weeks 2,4,6,8,10,12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale
  Baseline | 12.2 (5.45) | 12 (2.75)
  Week 2 | 10 (6.16) | 12.2 (1.32)
  Week 4 | 11.6 (5.08) | 13.2 (3.12)
  Week 6 | 11.8 (4.12) | 12 (1.79)
  Week 8 | 10.4 (3.93) | 9.8 (4.99)
  Week 10 | 11.6 (4.03) | 12.8 (1.17)
  Week 12 | 12.4 (4.41) | 12 (3.03)

5. Secondary Outcome: Change in Diagnostic Analysis of Nonverbal Activity-2 ADULT FACIAL EXPRESSIONS: (DANVA2-AF)
Description: This scale is shown to be sensitive to change in adults with autism, and related to amygdala function. Higher scores mean a better outcome.A clinical tool measuring emotion recognition through facial expression, voice and posture.
  1. Child faces 2 (range 0 - 100, higher values reflecting higher % of errors)
  2. Adult faces 2 (range 0 - 100, higher values reflecting higher % of errors)
  3. Child paralanguage 2 (range 0 - 100, higher values reflecting higher % of errors)
  4. Adult paralanguage 2 (range 0 - 100, higher values reflecting higher % of errors) Errors are counted and organized by pre-determined affect and intensity. Subtests considered separately.
Time Frame: baseline, weeks 2,4,6,8,10,12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Milnacipran | Placebo
Number analyzed (Participants) | 5 | 5
score on a scale
  Baseline | 16.5 (2.18) | 18.5 (3.5)
  Week 2 | 19.25 (1.48) | 19 (2.2)
  Week 4 | 19.6 (3.5) | 19.6 (2.06)
  Week 6 | 19.4 (4.08) | 20 (1.41)
  Week 8 | 17 (3.74) | 19.2 (1.94)
  Week 10 | 17.25 (3.77) | 20 (0.81)
  Week 12 | 18 (2.83) | 18.8 (2.78)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline to endpoint, for 12 weeks total.
Description: By definition, serious Adverse Events includes adverse events that result in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect.
Arm/Group | Milnacipran | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Milnacipran (N=5) | Placebo (N=5)
Fatigue (General disorders) | 2 | 0
Headache (General disorders) | 2 | 2
Nightmares (General disorders) | 0 | 2
Weight loss (General disorders) | 1 | 0
Abdominal Cramping (General disorders) | 1 | 0
Anal Fissure (Gastrointestinal disorders) | 1 | 0
Dizziness (General disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Gum Pain (General disorders) | 1 | 0
Hemorrhoids (General disorders) | 1 | 0
Insomnia (General disorders) | 1 | 0
Lethargy (General disorders) | 0 | 1
Lightheadedness (General disorders) | 0 | 1
Menstrual Cramps (General disorders) | 0 | 1
Nausea (General disorders) | 1 | 0
Sleep Disruption (General disorders) | 1 | 0
Stomachache (General disorders) | 0 | 1
Somnolence (General disorders) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 3 | 1
Vomiting (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No